CLINICAL TRIAL: NCT05227209
Title: A 12-Month Open-label Extension Study to Evaluate the Long-term Safety, Tolerability, and Effectiveness of SEP-4199 Controlled Release (CR) for the Treatment of Major Depressive Episode Associated With Bipolar I Disorder (Bipolar I Depression)
Brief Title: A Clinical Trial to Determine the Long-term Safety and Tolerability of an Investigational Drug in People With Major Depressive Episode Associated With Bipolar I Disorder (Bipolar I Depression).
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decided not to move forward with further accrual.
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEP380-303; 2021-002108-11 (EudraCT Number); jRCT2031220302 (Registry Identifier: Japan Registry for Clinical Trials)
Record Dates: First submitted 2022-01-27; First posted 2022-02-07 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Depressive Episodes, Bipolar I Depression
Keywords: Depression, Depressive episode, Bipolar, Bipolar 1, Bipolar 1 depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: This is a 12-month open-label safety extension study to evaluate the long-term safety, tolerability, and effectiveness of SEP-4199 CR 200-400 mg/day in the treatment of subjects with bipolar I depression who previously completed a lead-in study of SEP-4199 CR.The study will consist of a 12-month open-label flexible-dose treatment period, and a safety follow-up period
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SEP-4199 CR (Experimental): SEP-4199 CR either 200 mg (one 200 mg tablet) or 400 mg (two 200 mg tablets) once daily during open-label flexible-dose treatment period.
  Interventions: Drug: SEP-4199 CR

INTERVENTIONS:
Drug: SEP-4199 CR — SEP-4199 CR either 200 mg (one 200 mg tablet) or 400 mg (two 200 mg tablets) once daily

SUMMARY:
This is a clinical trial to determine the long-term safety and tolerability of an investigational drug in people with Major Depressive Episode Associated with Bipolar I Disorder (Bipolar I Depression). Participants in the study will receive the drug being studied. This study is accepting male and female participants between 18 and 65 years old who have completed Study SEP380-301. This study will be conducted in approximately 90 study centers worldwide. The treatment duration for this study is one (1) year.

DETAILED DESCRIPTION:
This is a 12-month open-label safety extension study to evaluate the long-term safety, tolerability, and effectiveness of SEP-4199 CR 200-400 mg/day in the treatment of subjects with bipolar I depression who previously completed a lead-in study of SEP-4199 CR.

The study will consist of a 12-month open-label flexible-dose treatment period, and a safety follow-up period. There are 15 scheduled visits, including a Baseline visit, 13 visits during the open-label treatment period, and 1 safety follow-up visit 7 (± 2) days after the last dose of study drug. If necessary, subjects may return to the clinic at anytime for an unscheduled visit

ELIGIBILITY:
Inclusion Criteria:

* Subject provides written informed consent and is willing and able to comply with the protocol in the opinion of the Investigator.
* Subject has completed 6 weeks of double-blind treatment and all scheduled assessments from Visit 6/EOT (Day 42) of the lead-in study of SEP-4199 CR.
* Subject is medically appropriate for long-term open-label treatment with SEP-4199 CR in the opinion of the Investigator.
* Female subjects of childbearing potential must agree to use effective and reliable contraception throughout the study and for at least 30 days after the last dose of study drug has been taken. In the Investigator's judgment, the subject will adhere to this requirement.
* Male subjects agree to avoid fathering a child and to use effective methods of birth control throughout the study and until at least 90 days after the last study drug administration.

Exclusion Criteria:

* Subject is at high risk of non-compliance in the opinion of the Investigator.
* Subject plans to initiate treatment with a prohibited psychotropic medication during the study.
* Subject plans to initiate treatment with transcranial magnetic stimulation (TMS), electroconvulsive therapy (ECT), vagus nerve stimulation (VNS), or deep brain stimulation (DBS) during the study.
* Subject experienced a moderate or severe hyperprolactinemia-related AESI in the lead-in study of SEP-4199 CR.
* Subject will require treatment with a drug that is associated with increases in QTc interval.
* Subject had any of the following at Visit 6/EOT (Day 42) of the lead-in study of SEP-4199 CR based on machine reading:
* increase in QTcF interval of ≥ 30 msec AND a QTcF interval ≥ 480 msec, from baseline of the lead-in study of SEP-4199 CR AND a QTCF interval ≥ 480msec
* increase in QTcF interval ≥ 60 msec, from baseline of the lead-in study of SEP-4199 CR
* QTcF interval ≥ 500 msec
* treatment-emergent clinically significant ECG abnormality.
* Subject is considered by the Investigator to be at imminent risk of suicide or injury to self or others, has a MADRS item 10 (suicidal ideation) score ≥ 4, or answers "yes" to "suicidal ideation" item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) on the C-SSRS assessment at Visit 6/EOT (Day 42) of the lead-in study of SEP-4199 CR.
* Female subject of childbearing potential, has a positive urine pregnancy test at Visit 6/EOT (Day 42) of the lead-in study of SEP-4199 CR or plans to become pregnant during the current study.
* Subject tests positive for any drug of abuse or cannabis at Visit 6/EOT (Day 42) of the lead-in study of SEP-4199 CR

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CNS Medical Director, Study Chair — Sumitomo Pharma America, Inc.
Locations (69):
- United States (25):
  - University of Alabama at Birmingham Huntsville Regional Medical Campus, Huntsville, Alabama
  - Advanced Research Center, Inc., Anaheim, California
  - Sun Valley Research Center, Imperial, California
  - Clinical innovations, Inc., Riverside, California
  - Collaborative Neuroscience Research, LLC, Torrance, California
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Premier Clinical Research Institute, Inc, Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Atlanta Behavioral Research, LLC, Atlanta, Georgia
  - Psych Atlanta, P.C., Marietta, Georgia
  - AMR Conventions Research, Warrenville, Illinois
  - St. Charles Psychiatric Associates / Midwest Research Group, Saint Charles, Missouri
  - Alivation Research, LLC, Lincoln, Nebraska
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Finger Lakes Clinical Research, Rochester, New York
  - Richmond Behavioral Associates ERG Clinical Research - New York PLLC, Staten Island, New York
  - New Hope Clinical Research, Charlotte, North Carolina
  - Quest Therapeutics of Avon Lake, Avon Lake, Ohio
  - Neuro-Behavioral Clinical Research, Inc, North Canton, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Lehigh Center for Clinical Research, LLC, Allentown, Pennsylvania
  - Community Clinical Research, Inc., Austin, Texas
  - UTHealth Science Center at Houston, Houston, Texas
  - Family Psychiatry of The Woodlands, The Woodlands, Texas
- Bulgaria (10):
  - State Psychiatric Hospital - Kardzhali First Women Department Third Men Department, Kardzhali
  - Medical Center Mentalcare OOD, Plovdiv
  - Mental Health Center- Ruse EOOD Men Department for treatment of persons with acute psychotic disorders; Women Department for treatment of persons with acute psychotic disorders; Department "Daily stationary", Rousse
  - Mental Health Center - Sofia EOOD, Sofia
  - Medical Center Sveti Naum EOOD, Sofia
  - DCC St. Vrach and St. St. Kuzma and Damian OOD, Sofia
  - Medical Center Hera EOOD, Sofia
  - Medical Center Intermedica OOD, Sofia
  - State Psychiatric Hospital - s. Tsarev brod First Department for Active Treatment - Men Second Department for Active Treatment - Men Women Department - Rehabilitation Sector Women Department - Acute Sector, Tsarevo
  - DCC Mladost-M Varna OOD, Varna
- Japan (34):
  - Hiro Mental Clinic, Fukuoka, Fukuoka
  - Shinseikai Kaku Mental Clinic, Fukuoka, Fukuoka
  - Mental Clinic Sakurazaka, Fukuoka, Fukuoka
  - Hatakeyama Clinic, Kitakyushu, Fukuoka
  - Someikai Kanagami Clinic, Kitakyushu-shi, Fukuoka
  - Kokura Mental Clinic, Kitakyushu-shi, Fukuoka
  - Hirota Clinic, Kurume-shi, Fukuoka
  - Shiranui Hospital, Omuta-shi, Fukuoka
  - Jisenkai Nanko Psychiatric Institute, Shirakawa-shi, Fukushima
  - Teine Keijinkai Hospital, Sapporo, Hokkaido
  - Tatsuta Clinic, Kobe, Hyōgo
  - Cerisier Heart Clinic, Kagoshima, Kagoshima-ken
  - Musashikosugi J Kokorono Clinic, Kawasaki, Kanagawa
  - Yutaka Clinic, Sagamihara-shi, Kanagawa
  - Azamino Mental Clinic, Yokohama, Kanagawa
  - Yamatenomori Kokorono Clinic, Yokohama, Kanagawa
  - Satokai Yuge Hospital, Kumamoto, Kumamoto
  - Shiroma Clinic, Urasoe-shi, Okinawa
  - Rainbow & Sea Hospital, Karatsu-shi, Saga-ken
  - Juntendo University Hospital, Bunkyō City, Tokyo-To
  - Senzoku Psychosomatic Clinic, Meguro-ku, Tokyo-To
  - Minami-Aoyama Antique Street Clinic, Minatoku, Tokyo-To
  - Heart Care Ginga Clinic, Nakano, Tokyo-To
  - Sangenjaya Nakamura Mental Clinic, Setagaya-Ku, Tokyo-To
  - Sangenjaya Neurology- Psychosomatic Clinic, Setagaya-Ku, Tokyo-To
  - Japanese Red Cross Medical Center, Shibuya-ku, Tokyo-To
  - Maynds Tower Mental Clinic, Shibuya-ku, Tokyo-To
  - Sangubashi Kokorono Clinic, Shibuya-ku, Tokyo-To
  - Etoh Mental Clinic, Shinagawa-ku, Tokyo-To
  - Tamaki Clinic, Shinjuku-ku, Tokyo-To
  - Himorogi Psychiatric Institute, Shinjuku-Ku, Tokyo-To
  - Uguisudani Mental Clinic, Taito-ku, Tokyo-To
  - Ohwa Mental Clinic, Toshima-ku, Tokyo-To
  - Kitaikebukuro Kokoro No Clinic, Toshima-ku, Tokyo-To

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study may be made available upon request via theVivli Center for Global Clinical Reserach Data site
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD will be made available upon request within 12 months of posting the study results on ct.gov.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://vivli.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study will consist of a 12-month open-label flexible-dose treatment period, and a safety follow-up period.All subjects will initiate treatment with SEP-4199 CR 200 mg/day. Study medication dose may be increased to 400 mg/day is at the Month 1 visit, based on the Investigator's judgment. The dose may be decreased to a minimum of 200 mg/day at any time thereafter for tolerability.
Period: Overall Study
Arm/Group | SEP-4199 CR
Started | 64
Completed | 9
Not Completed | 55
Not completed — Adverse Event | 11
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 7
Not completed — Other Early Termination Reason (Not Listed on CRF) | 36

BASELINE CHARACTERISTICS:
Arm/Group | SEP-4199 CR
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.8 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 59
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 20
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 43
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Experienced Adverse Events in Study
Description: Incidence of adverse events
Time Frame: 12 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | SEP-4199 CR
Number analyzed (Participants) | 64
Participants | 39

2. Primary Outcome: Number of Subjects Who Discontinued Due to Adverse Events
Description: Incidence of adverse events leading to discontinuation
Time Frame: 12 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | SEP-4199 CR
Number analyzed (Participants) | 64
Participants | 9

3. Primary Outcome: Number of Subjects Who Experienced Serious Adverse Events in Study
Description: Incidence of Serious Adverse Events
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | SEP-4199 CR
Number analyzed (Participants) | 64
Participants | 3

4. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Total Score - Change From Baseline
Description: Open Label (OL) Month 12 (LOCF) is defined as the last non-missing post-OL Baseline measurement up to and including the OL Month 12 measurement and within 9 days post the last dose of open-label extension study medication. The MADRS is a clinician-rated assessment of the subject's level of depression. The measure contains 10 items that measure apparent and reported sadness, inner tension, reduced sleep and appetite, difficulty concentrating, lassitude, inability to feel, and pessimistic and suicidal thoughts. Each item is scored in a range of 0 to 6 points and total score range is of 0 to 60 with higher scores indicating increased depressive symptoms.Individual items are then summed to determine total score.
Time Frame: 12 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SEP-4199 CR
Number analyzed (Participants) | 64
score on a scale | -6 (12.54)

5. Secondary Outcome: Clinical Global Impression Bipolar Version (CGI-BP-S) Depression Score - Change From Baseline
Description: Open Label (OL) Month 12 (LOCF) is defined as the last non-missing post-OL Baseline measurement up to and including the OL Month 12 measurement and within 9 days post the last dose of open-label extension study medication.The Clinical Global Impression Bipolar Version (CGI-BP-S) scale is a clinician-rated assessment of the subject's current illness state on a 7-point scale, where a higher score is associated with greater illness severity. Depression Score is one the individual item on CGI-BP-S Scale.The CGI-BP-S depression score takes one of the following values: 1 (normal, not at all ill), 2 (borderline mentally ill), 3 (mildly ill), 4 (moderately ill), 5 (markedly ill), 6 (severely ill), 7 (among the most extremely ill patients).
Time Frame: 12 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SEP-4199 CR
Number analyzed (Participants) | 64
score on a scale | -0.8 (1.34)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | SEP-4199 CR
All-Cause Mortality (participants affected / at risk) | 0/64
Serious Adverse Events (participants affected / at risk) | 3/64
Other Adverse Events (participants affected / at risk) | 39/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SEP-4199 CR (N=64)
Sarcoidosis (Immune system disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SEP-4199 CR (N=64)
Nasopharyngitis (Infections and infestations) | 5 (6)
Hyperprolactinaemia (Endocrine disorders) | 6 (6)
Depression (Psychiatric disorders) | 4 (6)
Insomnia (Psychiatric disorders) | 4 (4)
Headache (Nervous system disorders) | 4 (4)
Blood prolactin increased (Investigations) | 20 (20)
Weight increased (Investigations) | 5 (5)
Electrocardiogram QT prolonged (Investigations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.

DOCUMENTS (2):
  • Study Protocol (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/09/NCT05227209/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-25): https://cdn.clinicaltrials.gov/large-docs/09/NCT05227209/SAP_001.pdf